CLINICAL TRIAL: NCT04466358
Title: Comparison of CLOSE Guided and High Density Mapping Guided Catheter Ablation of Paroxysmal Atrial Fibrillation
Brief Title: CLOSE Versus High Density Mapping Guided Catheter Ablation of Paroxysmal Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Matevz Jan, Principal investigator, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLOSEVSHD
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Pulmonary Vein Isolation
Keywords: pulmonary vein isolation; paroxysmal atrial fibrillation; high density mapping
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified CLOSE protocol (Experimental): Width antral circumferential pulmonary vein isolation guided according to CLOSE protocol, confirmed with multipolar circular mapping catheter.
  Interventions: Procedure: Modified CLOSE protocol
- High density mapping guided pulmonary vein isolation (Active Comparator): Width antral circumferential pulmonary vein isolation guided according to CLOSE protocol and confirmed with high density mapping of each pulmonary vein antrum, with additional ablation lesions at sites of gap or dormant conduction.
  Interventions: Procedure: High density mapping guided pulmonary vein isolation

INTERVENTIONS:
Procedure: Modified CLOSE protocol — Modified CLOSE protocol guided isolation of pulmonary veins.
  Arms: Modified CLOSE protocol
Procedure: High density mapping guided pulmonary vein isolation — Modified CLOSE protocol guided isolation of pulmonary veins with additional ablations at sites of gaps or dormant conduction as evidenced by high density mapping of pulmonary vein antra.
  Arms: High density mapping guided pulmonary vein isolation

SUMMARY:
The aim of this study is to compare two methods of catheter ablation for treatment of paroxysmal atrial fibrillation (AF). The first method being a modified CLOSE protocol used for the control group and the second high density mapping guided isolation of pulmonary veins used for the interventional group. Comparison will be made according to clinical parameters and also durability of pulmonary vein isolation.

DETAILED DESCRIPTION:
CLOSE protocol is among the latest methods of catheter ablation of AF. According to this protocol, ablations are guided by ablation index, which takes into account ablation time, the contact force and power supplied by the ablation catheter. In this protocol the distance between individual ablation lesions is less than 6 millimeters (mm), thus ensuring the continuity of the ablation line around the pulmonary veins. After ablation, the electrical isolation of pulmonary veins (entry and exit block) is checked with a multi-electrode circumferential catheter. The electrical inactivity of the ablation line itself is thus checked indirectly via the conduction block. According to recent studies, the success rate of catheter ablation with this protocol after one procedure at one year is approximately 90%. Investigators believe that the presence of electrical activity within the ablation line, which does not translate into and out of the pulmonary veins during the procedure and is not detected by the currently used mapping technique, significantly affects the subsequent clinical success of the procedure. Investigators assume that high-resolution mapping of the ablation line would identify areas of electrical activity within the ablation line (dormant conduction) and that the ablation of these areas during the first procedure would significantly affect both the long-term isolation of the pulmonary veins and the clinical success of the procedure.

The aim of this study is to compare long-term clinical efficacy and efficacy of pulmonary vein isolation of two different methods of catheter ablation for treatment of AF. Participants will be randomised into two groups. In the first group isolation of pulmonary veins will be performed following a modified CLOSE protocol, the isolation will be checked with multipolar circumferential catheter. In the second group the ablation will be performed with the same method but the isolation of pulmonary veins will be checked with high-resolution mapping looking for dormant conduction in the pulmonary vein antra.

Hypothesis:

investigators expect that the incidence of the recurrence od AF in the high resolution mapping group will be lower during clinical follow-up. Investigators also expect that durable pulmonary vein isolation will be present in higher proportion of participants where high resolution mapping was performed.

Study protocol:

Participants will be randomized 1:1 into two groups:

1. Wide antral circumferential isolation of the pulmonary veins following modified CLOSE protocol (1) - ablation index at the posterior side 400, at the anterior side 550; distance between lesions <6 mm. 30 minutes after the completion of the ablation line, the isolation of the pulmonary veins is checked by inserting multipolar circular catheter into each pulmonary vein. In case of electrical activity ablation is added to close the gap in the line until pulmonary veins are electrically isolated.
2. Wide antral circumferential isolation of the pulmonary veins following modified CLOSE protocol (1) - ablation index at the posterior side 400, at the anterior side 550; distance between lesions <6 mm. 30 minutes after the completion of the ablation line, the isolation of the pulmonary veins is checked by inserting multipolar circular catheter into each pulmonary vein. Additionally a high density map is created with the multipolar catheter with at least 1000 mapping points for each pulmonary antrum. Signals considered to represent gaps in the line: multicomponent intracardiac electrograms consisting of at least three baseline deviations and/or conduction from vein to the atrium during pacing beyond ablation line (10 milliAmpers, 1 millisecond) and/or voltage amplitude inside the ablation line above 0.1 milliVolts. If intracardiac signals after added ablation on the line persist after additional ablations this region is not considered a gap in the line. The area of the gap is ablated until electric inactivity of the pulmonary vein antrum as evidenced with high density remapping.

Investigators will record the characteristics of the areas where gaps will be recorded: inappropriate drop in impedance during ablation (below 10 Ohms), the parameters of the contact force of the ablation catheter tip during ablation, interlesion distance, characteristics of unipolar recordings of intracardiac electrograms from the tip of the ablation catheter and others.

Twelve (12) months after the procedure, all participants (even without proven atrial tachyarrhythmia) will undergo a re-intervention to check electrical isolation of the pulmonary veins and pulmonary vein antra with a multi-electrode mapping catheter and high density mapping. In case of proven re-isolation of the pulmonary veins or their antra, investigators will find the location of the gap in the ablation line and add additional ablation at this location until electrical isolation will be achieved.

Follow-up:

All participants will have continuous electrocardiogram (ECG) monitoring for at least 12 hours after the procedure.

On the day after the procedure following examinations will be performed:

* 12-lead ECG,
* transthoracic ultrasound of the pericardium,

All participants will be monitored clinically for at least 12 months after the procedure:

After 3 months of blanking period, participants will come for the first outpatient examination in outpatient clinic of the University Medical Center in Ljubljana. This will be followed by a second outpatient examination after 6 months and a third outpatient examination after 12 months of intervention. In case of palpitations participants will be instructed to come to an earlier examination.

Clinical efficacy of the procedure will be defined as absence of AF episodes longer than 30 seconds detected by 24-hour ECG monitoring. Additionally, episodes of AF detected with event monitors and symptom driven 12-lead ECG recordings will be considered a recurrence.

On the first and second clinical follow-up (3, 6 months) the following examinations will be performed:

* history taking and clinical examination,
* 12-lead ECG recording,
* 24-hour Holter ECG,
* 1 week event monitor with daily 2 minute ECG recordings that will be sent to the investigator.

On the third clinical follow-up (12 months) the following examinations will be performed:

* history taking and clinical examination,
* 12-lead ECG recording,
* 24-hour Holter ECG,
* 1 week event monitor with daily 2 minute ECG recordings that will be sent to the investigator,
* transthoracic ultrasound of the heart.

Medical management: Antiarrhythmic drug (AAD) and anticoagulation (AC) management will be directed by the referring physician. Anticoagulation is continued post-procedurally for at least three months. This continuation of ADDs and AC will be controled by the referring physician and a predefined protocol for discontinuation will not be provided. Subsequent interventions including repeat catheter ablation will be directed by the referring physician and recorded.

ELIGIBILITY:
Inclusion Criteria:

* electrocardiographic evidence of paroxysmal AF in the last six months,
* unsuccessful treatment with antiarrhythmic drugs or highly symptomatic arrhythmia episodes (EHRA 3 and 4).

Exclusion Criteria:

* age over 80 years,
* greatly enlarged left atrium (ultrasound parasternal diameter more than 50 mm),
* life expectancy less than one year,
* acute life-threatening disease,
* previous heart surgery,
* severe left or right ventricular dysfunction (LVEF equal or less than 35 %),
* severe valve failure,
* presence of a clot in the left atrium,
* previous atrial fibrillation ablation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Recurrence of atrial fibrillation | 3-12 months
  Atrial fibrillation recorded with 12-lead ECG, event monitor or a 30 seconds episode recorded with Holter ECG.
Durability of pulmonary vein isolation | 12 months
  Presence of gaps in the circumferential ablation line (reconduction of pulmonary veins) as evidenced at predefined remapping procedure.

SECONDARY OUTCOMES:
Characteristics of gaps in ablation lines | 0-12 months
  Characteristics of electrograms and ablation lesions in the areas where gaps in the ablation line will be discovered acutely during high density mapping at index procedure. Also, characteristics of electrograms and ablation lesions in the areas where gaps will be discovered at a remote re-mapping procedure at 12 months after the index procedure

OTHER OUTCOMES:
Adverse events | 0-1 month
  During and after the procedure and at clinical follow-ups, any serious adverse event will be recorded. Significant adverse events will be defined as all events that endanger the participant's health or prolong hospitalization, or require intervention:
  * Death in hospital
  * Pericardial effusion resulting in tamponade
  * Cerebral insult
  * Pneumonia
  * Phrenic nerve injury
  * Esophageal perforation
  * Cardiac arrest
  * Complete atrioventricular block
  * Vascular intervention and / or surgery
  * Transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Jernej Stublar, MSE, Study Director — University Medical Centre Ljubljana; Bor Antolic, MD, PhD, Study Chair — University Medical Centre Ljubljana
Locations (1):
- UMC Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Phlips T, Taghji P, El Haddad M, Wolf M, Knecht S, Vandekerckhove Y, Tavernier R, Duytschaever M. Improving procedural and one-year outcome after contact force-guided pulmonary vein isolation: the role of interlesion distance, ablation index, and contact force variability in the 'CLOSE'-protocol. Europace. 2018 Nov 1;20(FI_3):f419-f427. doi: 10.1093/europace/eux376. PMID 29315411
- [Background] Taghji P, El Haddad M, Phlips T, Wolf M, Knecht S, Vandekerckhove Y, Tavernier R, Nakagawa H, Duytschaever M. Evaluation of a Strategy Aiming to Enclose the Pulmonary Veins With Contiguous and Optimized Radiofrequency Lesions in Paroxysmal Atrial Fibrillation: A Pilot Study. JACC Clin Electrophysiol. 2018 Jan;4(1):99-108. doi: 10.1016/j.jacep.2017.06.023. Epub 2017 Sep 27. PMID 29600792
- [Background] Duytschaever M, De Pooter J, Demolder A, El Haddad M, Phlips T, Strisciuglio T, Debonnaire P, Wolf M, Vandekerckhove Y, Knecht S, Tavernier R. Long-term impact of catheter ablation on arrhythmia burden in low-risk patients with paroxysmal atrial fibrillation: The CLOSE to CURE study. Heart Rhythm. 2020 Apr;17(4):535-543. doi: 10.1016/j.hrthm.2019.11.004. Epub 2019 Nov 9. PMID 31707159
- [Background] Meissner A, Maagh P, Christoph A, Oernek A, Plehn G. Pulmonary vein potential mapping in atrial fibrillation with high density and standard spiral (lasso) catheters: A comparative study. J Arrhythm. 2017 Jun;33(3):192-200. doi: 10.1016/j.joa.2016.10.562. Epub 2016 Nov 25. PMID 28607614
- [Background] Segerson NM, Lynch B, Mozes J, Marks MM, Noonan DK, Gordon D, Jais P, Daccarett M. High-density mapping and ablation of concealed low-voltage activity within pulmonary vein antra results in improved freedom from atrial fibrillation compared to pulmonary vein isolation alone. Heart Rhythm. 2018 Aug;15(8):1158-1164. doi: 10.1016/j.hrthm.2018.04.035. Epub 2018 May 3. PMID 29729399
- [Derived] Kajdic N, Kalinsek TP, Antolic B, Zizek D, Stublar J, Demsar J, Kuhelj D, Jan M. Impact of High-Density Mapping on Pulmonary Vein Isolation Durability: A Randomized, Single-Center Study. Pacing Clin Electrophysiol. 2025 Jun;48(6):587-597. doi: 10.1111/pace.15196. Epub 2025 May 6. PMID 40326295